CLINICAL TRIAL: NCT06583148
Title: Assessing the Effectiveness of a Smoke-Free Home Program in Tribal Communities
Brief Title: A Smoke-Free Home Intervention in Tribal Communities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Michelle C. Kegler, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00006459; NCI-2024-06174 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00006459 (Other: Emory University Hospital/Winship Cancer Institute); RSPH6261-24 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH); R01CA268024 (NIH)
Record Dates: First submitted 2024-08-14; First posted 2024-09-03 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Tobacco-Related Carcinoma
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Smoking Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Randomization will be supervised by the study statistician and data collection staff will be blind to group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (smoke-free home program) (Experimental): Participants receive the smoke-free home program, consisting of mailed educational information about smoke-free homes at enrollment and in weeks 4 and 6, and attend one coaching call in week 2.
  Interventions: Behavioral: Smoking Cessation Intervention; Other: Survey Administration
- Group II (waitlist control) (Active Comparator): Participants receive usual care on study. Participants may optionally receive the smoke-free home program following the 6 months follow-up.
  Interventions: Other: Best Practice; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Group II (waitlist control)
Behavioral: Smoking Cessation Intervention — Receive the smoke-free home program
  Other Names: Smoking and Tobacco Use Cessation Interventions
  Arms: Group I (smoke-free home program)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates a smoke-free home intervention for reducing exposure to secondhand smoke from commercial tobacco in homes of participants who live in rural tribal communities. Smoke-free homes are an innovative and relatively untapped strategy for cancer prevention in rural tribal communities. Smoke-free policies, including those that target homes, can reduce exposure to secondhand smoke and support smoking cessation. Rural and racial/ethnic inequities intersect to increase tobacco-related harms among Indigenous populations. A smoke-free home program may improve the health of the household as well as impact smoking behavior among the family unit by reducing secondhand smoke exposure.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the effectiveness of a smoke-free homes intervention for tribal communities.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP I: Participants receive the smoke-free home program, consisting of mailed educational information about smoke-free homes at enrollment and in weeks 4 and 6, and attend one coaching call in week 2.

GROUP II: Participants receive usual care on study. Participants may optionally receive the smoke-free home program following the 6 months follow-up.

After completion of study intervention, participants are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Self-report as being a smoker or living with a smoker
* Indicate that they do not reside in a smoke-free home
* Identify as living in an American Indian household

Exclusion Criteria:

* Children under the age of 18 will not be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 575 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Self-Reported Smoke-Free Home | At 3 and 6 months
  Which statement best describes rules about smoking inside your home? There are no rules about smoking inside your home? Smoking is not allowed anywhere inside your home? Smoking is allowed in some places or at some times in your home? Smoking is allowed anywhere inside your home? Those answering that smoking is not allowed anywhere inside their home are classified as having a smoke-free home. It will be self-reported & measured using air nicotine monitor from a subset of 20% participants to assess validity of the self-report, adjusting for possible traditional uses of tobacco and use of electronic cigarettes. Receiver-operator curve analysis to determine the optimal thresholds for a smoke-free home & complete case data, two-level logistic multilevel models accounting for nesting of participants in tribal communities with group assignment predicting a binary smoke-free home status (full ban/no full ban).

SECONDARY OUTCOMES:
Smoke-Free Vehicles Assessed Via Telephone Interview | At 3 and 6 months
  Smoke-Free Vehicles will be assessed via telephone interview using a measure adapted from the Centers for Disease Control and Prevention (CDC)'s National Adult Tobacco Survey, 2009-2010. What about smoking cigarettes in your vehicle(s) (including cars, SUVs, and trucks) - would you say: There are no rules about smoking in the vehicle(s), smoking is sometimes allowed in the/some vehicle(s), smoking is never allowed in the/any vehicle, no car, don't know. Those answering smoking is never allowed in the/any vehicle are classified as having a smoke-free vehicle rule. We will use 3-level logistic growth curve models using Statistical Analysis System (SAS) procedure (PROC) Bayesian Generalized Linear Mixed Modeling (BGLIMM) to model all of the collected data. Data cleaning, descriptive analyses, as well as bivariate and multilevel modeling, will be conducted using Statistical Analysis System (SAS) version 9.4. Mediation analyses will be conducted in Mplus statistical software version 8.5.
Secondhand Smoke (SHS) Exposure In The Home Assessed via Telephone Interview | At 3 and 6 months
  SHS exposure in the home will be assessed via telephone interview using a measure adapted from the Centers for Disease Control and Prevention (CDC)'s National Youth Tobacco Survey, 2023. During the past 7 days, how many days have people smoked in your home in your presence? Response options 0 to 7. We will use 3-level logistic growth curve models using Statistical Analysis System (SAS) procedure (PROC) Bayesian Generalized Linear Mixed Modeling (BGLIMM) to model all of the collected data. Data cleaning, descriptive analyses, as well as bivariate and multilevel modeling will be conducted using Statistical Analysis System (SAS) 9.4. Mediation analyses will be conducted in Mplus statistical software version 8.5.
Number of Cigarettes Smoked In the Home | At 3 and 6 months
  Will use 3-level logistic growth curve models using Statistical Analysis System (SAS) procedure (PROC) Bayesian Generalized Linear Mixed Modeling (BGLIMM) to model all of the collected data. Data cleaning, descriptive analyses, as well as bivariate and multilevel modeling will be conducted using Statistical Analysis System (SAS) version 9.4. Mediation analyses will be conducted in Mplus statistical software version 8.5.
Public Support for Smoke-Free Tribal Housing Assessed Via Telephone Interview | At 3 and 6 months
  To what extent do you support or oppose a complete cigarette smoking ban in the following settings: tribally owned multi-unit housing. Response options include a range from 1 (strongly oppose) to 4 (strongly support).

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Kegler, DrPH, MPH, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States